CLINICAL TRIAL: NCT05524337
Title: The Effect of White Noise and Therapeutic Touch on Physiological Parameters, Pain and Comfort Level in Newborns During Heel Blood Collection: A Randomized Controlled Study
Brief Title: White Noise and Therapeutic Touch on Pain and Comfort Level in Newborns During Heel Lance
Acronym: noisetouch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gülçin Özalp Gerçeker, Assoc. Prof., Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 6943 GOA
Record Dates: First submitted 2022-07-21; First posted 2022-09-01 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Pain, Acute; Newborn
MeSH Terms: conditions — Acute Pain | interventions — Therapeutic Touch

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- White noise group (Experimental): In the white noise group, it will be explained to the mother of the baby that the white noise sound to be used in the research will be used for pain relief. Dr. Harvery Karp's song "The Happiest Baby", consisting of intrauterine sounds only, will be used for white noise. The sound will be set to 45 db. The loudspeaker will be placed on the tip of the foot, approximately 30 cm from the newborns ear, five minutes before the procedure, and will be played to the baby during the procedure. 5 minutes without taking heel blood. Before, during the procedure and 5 minutes after the end of the procedure, this sound will be played to the baby and the data will be recorded by the observer.
  Interventions: Behavioral: white noise
- therapeutic touch group (Experimental): Therapeutic touch steps:
  1. Before the application, explaining the study and the intervention to be applied to the mother, obtaining the consent of the mother to participate in the study, and filling the introductory information form will be done at this stage.
  2. Immobile touching: Hands will be washed and warmed so that they do not disturb the baby. The researcher will support the babys back and hips with one hand, while holding the baby's chest and abdomen with the other hand. In the meantime, the nurse who will take the heel blood will start the process and continue to touch.
  3. Compassionate touch: While the practitioners hands are in the same position; He would caress for 1 minute, rest his hands for 30 seconds, then caress again for 1 minute, rest his hands for 30 seconds, and finally continued to caress for 2 minutes. The caressing process was completed by touching it with circular movements of 1 cm diameter in a clockwise direction every 10 seconds.
  Interventions: Behavioral: therapeutic touch
- therapeutic touch and white noise group (Experimental): the group where therapeutic touch and white noise will be applied together, after the family is informed about the procedure, white noise will be listened to 5 minutes before, during and 5 minutes after the heel blood collection, and therapeutic touch steps will be applied during this time. Meanwhile, the data will be recorded on the form by the observer.
  Interventions: Behavioral: white noise and therapeutic touch
- Control group (No Intervention): Non-pharmacological intervention will not be made for the baby in the control group,

INTERVENTIONS:
Behavioral: white noise — Dr. Harvery Karp's song "The Happiest Baby", consisting of intrauterine sounds only, will be used for white noise. The sound will be set to 45 db.
  Arms: White noise group
Behavioral: therapeutic touch — In the group where therapeutic touch will be applied, the heel blood collection procedure and the study will be explained to the family, and after the consent is obtained, the therapeutic touch will be applied to the baby 5 minutes before, during and after the procedure.
  Arms: therapeutic touch group
Behavioral: white noise and therapeutic touch — the group where therapeutic touch and white noise will be applied together, after the family is informed about the procedure, white noise will be listened to 5 minutes before, during and 5 minutes after the heel blood collection, and therapeutic touch steps will be applied during this time.
  Arms: therapeutic touch and white noise group

SUMMARY:
This randomized controlled study was planned to evaluate the effects of listening to white noise and therapeutic touch on physiological parameters, pain and comfort level during the heel blood collection procedure on infants who gave birth at 32 weeks and above and were given to their mothers in Atatürk Training and Research Hospital.

DETAILED DESCRIPTION:
Hypotheses

H1: Newborns who listen to white noise during heel blood collection feel less pain and have a higher comfort level. H2: Newborns who are treated with therapeutic touch during heel blood collection feel less pain and have a higher comfort level. H3: Newborns who listen to white noise and apply therapeutic touch during heel blood collection feel less pain and have a higher comfort level. H4: There is a difference between the pain and comfort levels of newborns in terms of group, group-time and time according to the intervention applied.

Methods

Mothers of newborns whose heel blood will be taken will be informed about the research. The mothers will be informed about the fact that heel blood collection is a routine practice, the data will be recorded by the nurse and 2 observers who take heel blood in the study, and they will also be informed about the white noise and therapeutic touch practices to be listened to, and their written consent will be obtained.

After obtaining informed written consent, it will be determined which group the newborn belongs to by stratified randomization. Stratified randomization was applied according to gender and week of birth.

A standard approach will be applied to all newborns. Standard approach; If the baby is asleep, the heel blood will be taken, he will be woken up, put on a denim bed, his upper extremities will be gently wrapped with a blanket, and the procedure will be performed by the nurse.

Babies to be included in the study in each group; Until 30 minutes before the start of the procedure, they will be in their beds, in the rest period, where they are not disturbed. All babies; 5 minutes before, during and up to 5 minutes after blood collection; Observational findings including heart rates, SpO2 values, pain and confort scores will be recorded in the data form. No additional care will be given to ensure physiological stability in all groups.

ELIGIBILITY:
Inclusion Criteria:

* Babies who are 32 weeks and older given to their mothers who were born healthy

Exclusion Criteria:

* Newborns 32 weeks and over
* Delivery of the newborn to the mother after birth
* no congenital anomalies or genetic disorders
* The newborn has passed the audiology test
* Obtaining consent form from parent

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-07-22 (Actual); Study Completion 2023-07-22 (Actual)

PRIMARY OUTCOMES:
Neonatal Infant Pain Scale (NIPS) | 5 minutes
  The Newborn Infant Pain Scale (NIPS) was developed by Lawrence et al. in 1993. Turkish validity and reliability were established by Akdovan in 1999 (Akdovan, 1999). Newborn infant pain scale, facial movements (0; relaxed, 1; restless), crying (0; no crying, 1; groaning, 2; loud crying), breathing (0; relaxed, 1; variable-irregular), arm (0 It is a likert-type scale consisting of 6 parameters: relaxed-free, 1; flexion-extension), leg (0; comfortable-free, 1; flexion-extension) and sleep-wake (0; sleeping-waking peaceful, 1; restless). . The assessment of pain is based on the total score.
The newborn comfort behavior scale | 5 minutes
  The newborn comfort behavior scale is a Likert type scale developed to evaluate the comfort needs, pain and distress of newborn babies. This scale was developed by Ambuel et al. (1992) to evaluate comfort, pain and stress in newborn babies receiving mechanical ventilator support in the intensive care unit (Ambuel et al., 1992). As a result of the application of this scale, a total score of 6-30 is reached. If the total score obtained as a result of the evaluation is between 9-13, it is emphasized that the baby is comfortable, if it is 14 and above, the baby's comfort level is low and additional interventions may be required to increase comfort.

SECONDARY OUTCOMES:
heart rate | 10 minutes
  Babies to be included in the study in each group; Until 30 minutes before the start of the procedure, they will be in their beds, in the rest period, where they are not disturbed. All babies; 5 minutes before, during and up to 5 minutes after blood collection. Heart rate will recorded.
oxygen saturation | 10 minutes
  Babies to be included in the study in each group; Until 30 minutes before the start of the procedure, they will be in their beds, in the rest period, where they are not disturbed. All babies; 5 minutes before, during and up to 5 minutes after blood collection. Oxygen saturation will recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Gülçin Özalp Gerçeker, Study Director — RN, PhD, Assoc. Prof.
Locations (1):
- Gülçin Özalp Gerçeker, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No